CLINICAL TRIAL: NCT05694910
Title: The Effect of Reiki on Fatigue, Vital Signs and Engraftment in Bone Marrow Transplant Patients
Brief Title: Reiki Effects on Bone Marrow Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, NURSEMIN UNAL, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 113
Record Dates: First submitted 2023-01-07; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Bone Marrow Transplant Complications; Fatigue; Vital Signs; Reiki
Keywords: Reiki; Fatigue; Vital signs; Engraftment; Bone marrow transplant patients
MeSH Terms: conditions — Fatigue | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patients and investigators knew which group they were assigned to. Only that outcome assessor did not know which patient was assigned to which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki Group (Experimental): Personal Information Form (PIF), Visual Analog Scale (VAS), and National Cancer Institute (NCI) -Common Terminology Criteria for Adverse Events (CTCAE) will be administered to the patients. Then vital signs and laboratory findings will be recorded. After the protests will be completed, the primary investigator with Reiki second degree will apply Reiki to the patients for 30 minutes. On the second day and the third day, 30 minutes distance Reiki will be applied to the patients. Post-tests will be applied to all patients after one week and vital signs and laboratory findings will be recorded.
  Interventions: Other: Reiki
- Control Group (No Intervention): Personal Information Form (PIF), Visual Analog Scale (VAS), and National Cancer Institute (NCI) -Common Terminology Criteria for Adverse Events (CTCAE) will be administered to the patients. Then vital signs and laboratory findings will be recorded. After a week, the posttest will be applied to the patients and vital signs and laboratory findings will be recorded.

INTERVENTIONS:
Other: Reiki — Reiki has based on the belief that disease occurs when an energy center is blocked, and that the energy is transmitted through touch. In distance Reiki, Reiki practitioners followed the traditional Usui Reiki protocol healing.
  Arms: Reiki Group

SUMMARY:
The aim of the study is to examine the effect of Reiki on fatigue, vital signs, and engraftment in bone marrow transplant patients.

DETAILED DESCRIPTION:
Cancer is a serious and chronic disease, the number of which is increasing rapidly in our country and in the world. Today, cancer accounts for 70% of all disease diagnoses and it is estimated that the number of new cancer cases will rise to 22 million in about twenty years.

Although hematopoietic stem cell transplantation is a promising treatment for remission and complete recovery in cancer patients, the symptoms after transplantation seriously affect the quality of life of individuals. In addition to psychosocial problems, patients experience serious physical problems such as suppression of the immune system and fatigue after transplantation. Energy therapies are widely used to provide general health and well-being and to reduce or relieve the symptoms of many chronic diseases. As a result of many studies on conditions such as fatigue, pain, and anxiety, it has been determined that Reiki energy has a positive effect. When we searched the literature, it was seen that there were not enough studies examining the fatigue, vital signs, and immune systems of bone marrow transplant patients.

This randomized controlled prospective study is conducted with bone marrow transplant patients between August 2022 to February 2023. The data of the study will collect using "Personal Information Form (PIF)", "Visual Analog Scale (VAS)", and "National Cancer Institute (NCI) -Common Terminology Criteria for Adverse Events (CTCAE)". Also, vital signs and laboratory findings will be recorded.

PIF, VAS, and CTCAE will be applied to the patients who meet the inclusion criteria. Patients will be randomized 1:1 into groups to the block randomization method. There are two arms in the study; Reiki (n=21) and control group (n=21). A second-degree Reiki practitioner will apply Reiki to the patients for 30 minutes. on the second day and the third day, 30 minutes distance Reiki will be applied to the patients. In the control group, nothing will be done. Post-tests will be applied to all patients after one week and vital signs and laboratory findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Not having a communication problem,
* Autologous bone marrow transplantation has been performed
* Willingness to participate in Reiki practice,
* To be competent to answer the data collection tools to be used in the research.
* Not using complementary practices (energy therapies) in the last six months.

Exclusion Criteria:

* Having a communication problem
* Application of allogeneic bone marrow transplantation
* Not being willing to engage in Reiki practice
* Reiki practitioner or instructor,
* Have received energy therapy sessions such as Reiki/Therapeutic touch/Healing touch in the last six months
* Application of bone marrow transplantation for hematological cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | Baseline
  There are questions to determine the soci-demographic features and the characteristics of the disease/treatment process.
Visual Analog Scale | Change from baseline Visual Analog Scale at one week
  It is a reliable and easily applicable scale used to measure the severity of pain in patients, accepted in the world literature. The scale, which was used to digitize the values that could not be measured numerically, was used to evaluate the pain intensity of the patients. A minimum of 0 and a maximum of 10 points can be obtained from the scale. In addition, high scores indicate increased pain intensity.
Fatigue | Change from fatigue level at a week
  Common Terminology Criteria for Adverse Events (CTCAE) define adverse events experienced by cancer patients. Patients are asked to number the level of fatigue from 0 to 10. As the score increases, the severity of fatigue also increases.
Engraftment | After one week
  Engraftment is when the transplanted stem cells grow and produce new blood cells at levels that can be counted in the bloodstream.
Change from Leukocyte values at a week | Change from Leukocyte values at a week
  They are the leading elements of the body's defense system.
Change from Hemoglobin values at a week | Change from Hemoglobin values at a week
  Hemoglobin is a substance found in red blood cells that makes it possible for the blood to carry oxygen throughout the body.
Change from Hematocrit values at a week | Change from Hematocrit values at a week
  Hematocrit refers to the ratio of the volume of red blood cells to the amount of circulating blood.
Change from Erythrocyte values at a week | Change from Erythrocyte values at a week
  The erythrocyte contains hemoglobin, which is involved in the transport of oxygen in the body.
Change from heart rate values at a week | Change from heart rate values at a week
  The number of times the heart beats per minute is the heart rate.
Change from systolic and diastolic blood pressure values at a week | Change from systolic and diastolic blood pressure values at a week
  Blood pressure is the pressure of the blood within the arteries of the circulatory system.
Change from body temperature values at a week | Change from body temperature values at a week
  Body temperature indicates the balance between the heat produced in the body and the heat consumed. A certain temperature is needed for the human body to continue its functions.
Change from respiratory rate values at a week | Change from respiratory rate values at a week
  At rest, the respiratory rate of an adult should be 12-20/min.
Change from oxygen saturation values at a week | Change from oxygen saturation values at a week
  Oxygen saturation refers to the oxygen saturation in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay BEKTAS AKPINAR, Principal Investigator — Ankara Medipol University
Locations (1):
- Nursemin Ünal, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simpson E, Dazzi F. Bone Marrow Transplantation 1957-2019. Front Immunol. 2019 Jun 5;10:1246. doi: 10.3389/fimmu.2019.01246. eCollection 2019. PMID 31231381
- [Background] Abo S, Denehy L, Ritchie D, Lin KY, Edbrooke L, McDonald C, Granger CL. People With Hematological Malignancies Treated With Bone Marrow Transplantation Have Improved Function, Quality of Life, and Fatigue Following Exercise Intervention: A Systematic Review and Meta-Analysis. Phys Ther. 2021 Aug 1;101(8):pzab130. doi: 10.1093/ptj/pzab130. PMID 33989413
- [Background] So WK, Dodgson J, Tai JW. Fatigue and quality of life among Chinese patients with hematologic malignancy after bone marrow transplantation. Cancer Nurs. 2003 Jun;26(3):211-9; quiz 220-1. doi: 10.1097/00002820-200306000-00006. PMID 12832954
- [Background] Cohen MZ, Rozmus CL, Mendoza TR, Padhye NS, Neumann J, Gning I, Aleman A, Giralt S, Cleeland CS. Symptoms and quality of life in diverse patients undergoing hematopoietic stem cell transplantation. J Pain Symptom Manage. 2012 Aug;44(2):168-80. doi: 10.1016/j.jpainsymman.2011.08.011. Epub 2012 Jun 13. PMID 22699091
- [Background] Smith MC, Reeder F, Daniel L, Baramee J, Hagman J. Outcomes of touch therapies during bone marrow transplant. Altern Ther Health Med. 2003 Jan-Feb;9(1):40-9. PMID 12564350
- [Background] Kelly DL, Syrjala K, Taylor M, Rentscher KE, Hashmi S, Wood WA, Jim H, Barata A, Flynn KE, Burns LJ, Shaw BE, Petersdorf E, Yero AC, Emmrich AD, Morris KE, Costanzo ES, Knight JM. Biobehavioral Research and Hematopoietic Stem Cell Transplantation: Expert Review from the Biobehavioral Research Special Interest Group of the American Society for Transplantation and Cellular Therapy. Transplant Cell Ther. 2021 Sep;27(9):747-757. doi: 10.1016/j.jtct.2021.06.007. Epub 2021 Jun 15. PMID 34139388
- [Background] Mische Lawson L, Glennon C, Fiscus V, Harrell V, Krause K, Moore AB, Smith K. Effects of Making Art and Listening to Music on Symptoms Related to Blood and Marrow Transplantation. Oncol Nurs Forum. 2016 Mar;43(2):E56-63. doi: 10.1188/16.ONF.E56-E63. PMID 26906139